CLINICAL TRIAL: NCT06757101
Title: Comparison of the Effects of Vojta and Bobath Treatment on Gait and Balance in Diplegic Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Unsa Baloch/ 01641
Record Dates: First submitted 2023-08-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: Cerebral palsy; Bobath Therapy; Vojta Therapy; balance; gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vojta Therapy group (Experimental): Vojta Therapy group for gait & balance
  Interventions: Other: Vojta Therapy
- Bobath Therapy group (Experimental): Bobath Therapy group for gait & balance
  Interventions: Other: Bobath Therapy
- Combined Vojta and Bobath therapy (Experimental): Combined Vojta and Bobath therapy for gait & balance
  Interventions: Other: Combined Vojta and Bobath Therapy

INTERVENTIONS:
Other: Vojta Therapy — Exercises will be performed in supine, lateral, decubitus and reflex crawling. Exercises will include Stretching's, ROMs Exercises, Stimulation of 10 different zones for locomotion & gentle pressure applied to stimulation areas. Frequency of exercises will be 2 times a week, duration 40 minutes per day.
  Arms: Vojta Therapy group
Other: Bobath Therapy — Exercises will be performed in supine, lateral, prone and standing position. Exercises includes stretching Exercises, ROMs, Quadruped imbalance exercise, Imbalance from the kneeling exercise, Cervant Knight exercise, Tandem walk, Kicking a ball, Step climbing, marching at one place with alternate foot Frequency of exercises will be 2 times a week, duration 40 minutes per day.
  Arms: Bobath Therapy group
Other: Combined Vojta and Bobath Therapy — Combined Vojta and Bobath exercises along with the conventional treatment. Frequency of exercises will be 2 times a week, duration 40 minutes per day.
  Arms: Combined Vojta and Bobath therapy

SUMMARY:
This study aims compare the effects of Vojta verses Bobath therapy on gait in children with diplegic cerebral palsy and to compare the effects of Vojta versus Bobath therapy on balance in children with diplegic cerebral palsy. The study will also determine the combined effects of Vojta and Bobath on gait and balance in children with diplegic cerebral palsy.

DETAILED DESCRIPTION:
The study may provide non-invasive and cost-effective treatment option in improving balance & gait in children with cerebral palsy. This can increase the child independence, confidence and quality of life. Additionally, this study may contribute to the development of evidence-based rehabilitation protocols, which can help guide clinical decision-making and treatment options. The study may provide insight into the feasibility and safety of combining Vojta and Bobath treatments, which can guide future research and practice in this area. Moreover, combination of treatments may have better outcomes as compared to the two individual techniques. The study aims compare the effects of Vojta verses Bobath therapy on gait in children with diplegic cerebral palsy and to compare the effects of Vojta versus Bobath therapy on balance in children with diplegic cerebral palsy. The study will also determine the combined effects of Vojta and Bobath on gait and balance in children with diplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of spastic diplegic cerebral palsy
* GMFCS level II & III
* Modified Ashworth score greater than 1+
* Age 3-8 Years
* Either gender
* Children capable of understanding and executing commands;
* Children who can adopt the orthostatic position necessary to assess balance & gait

Exclusion Criteria:

* Children with any other associated disease (DDH, any orthopedic complication)
* Children with mental retardation;
* Who cannot participate constantly in physical therapy sessions;
* Profound visual or hearing impairments;

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Gross Motor Functional Classification System (GMFCS) | 8 weeks
  The Gross Motor Functional Classification System (GMFCS) is the assessment tool to measure motor function in children with cerebral palsy. GMFCS is a five-level classification that differentiates children with Level I:Walks independently, Level II: Walks with limitations, Level III: Walks with hand- held mobility, Level IV: Self mobility with limitations, may use powered mobility & Level V: Transported in a manual wheelchair. The inter-rater reliability of GMFCS have a moderate agreement with a kappa (k) of 0.55 in children <2 years of age and excellent agreement with a kappa of 0.75 in children 2-12 years of age. This strong inter-rater reliability supports the use of the GMFCS as a classification of gross motor function in children ages 2-12 years.
Goniometer | 8 weeks
  The Goniometer measures the angle created at a joint by the adjacent bones of the body. Goniometer measurement represent the actual joint range of motion. There are multiple types of goniometer but universal goniometer is widely used in physiotherapy settings.
Paediatric Berg Balance Scale | 8 weeks
  The Paediatric Berg Balance Scale is used to assess functional balance skills in school-aged children. The scale consists of 14 items that scored from 0 points (lowest function) to 4 (highest function) with a maximum score of 56 points. Concurrent validity between Pediatric Balance Scale and GMFM at baseline (r=0.095), follow-up (r=0.44-0.87). Predictive validity of Pediatric validity and GMFM at follow-up (r=0.90-0.92) The test retest reliability is extremely high [(ICC3, 1=0.9987)].
Step Length | 8 weeks
  Step length is typically measured in centimeters (cm) or inches. Step length is used in clinical settings to assess gait abnormalities and has implications for rehabilitation. Adequate step length contributes to effective ambulation and helps maintain stability and momentum during walking.
Stride Length | 8 weeks
  Stride length is a key parameter in gait analysis that refers to the distance covered in one complete cycle of walking or running, specifically the distance between the initial contact point of one foot and the initial contact point of the same foot on the next step. Stride length is typically measured in units such as centimeters (cm) or inches. Stride length is critical in clinical assessments for identifying gait abnormalities.
Cadence | 8 weeks
  Cadence refers to the number of steps a person takes per unit of time, typically expressed as steps per minute (spm). It is a critical metric in gait analysis, providing insights into walking or running patterns and overall locomotion efficiency. A normal cadence (generally between 100 to 130 steps per minute for walking) is important for maintaining stability and rhythm during locomotion. Abnormal cadence can lead to increased fall risk and affect overall mobility.
Walking Base | 8 weeks
  Walking base, also known as base of support or stance width, refers to the distance between the feet when a person is walking. Specifically, it is the lateral distance between the heel centers of both feet during the walking cycle. A wider walking base indicates that the feet are positioned farther apart, while a narrower walking base means they are closer together. Walking base is typically measured in centimeters (cm).Walking base is a significant parameter in the assessment of gait and balance, providing insights into an individual's stability and mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Abrish Habib Abbasi, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Child Development Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No